CLINICAL TRIAL: NCT05677958
Title: Protein Intake in Patients With Colorectal or Lung Cancer During First Line Treatment With Chemo (Radio) - or Immunotherapy When Receiving a Low Volume, Energy Dense and High Protein Oral Nutritional Supplement: a Randomized, Controlled Study
Brief Title: Protein Intake in Patients With Colorectal or Lung Cancer When Receiving a Nutritional Supplement
Acronym: PROTEOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nutricia Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MPR16TA06151
Record Dates: First submitted 2022-11-23; First posted 2023-01-10 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Colorectal Cancer; Lung Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: Test group: receiving daily 2 servings of a low volume, energy dense and high protein oral nutritional supplement (ONS) Control group: not receiving any study product. These subjects will be receiving standard of care.
Masking Description: randomised controlled, open label, parallel-group, multi-centre and multicountry study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Active Comparator): 125 mL Fortimel/Nutridrink Compact Protein
  Interventions: Dietary Supplement: 125 mL Fortimel/Nutridrink Compact Protein
- Control group (No Intervention)

INTERVENTIONS:
Dietary Supplement: 125 mL Fortimel/Nutridrink Compact Protein — 125 mL Fortimel/Nutridrink Compact Protein®* two servings per day (300 kcal, 18 g protein per serving).
  Arms: Test group

SUMMARY:
The PROTEOS study is an randomized controlled, open label, parallel-group, multi-centre and multicounty interventional study to assess the acceptance and implementation of Compact Protein, a low volume, energy dense and high protein oral nutritional support in clinical practice according to the ESPEN guidelines in colorectal and lung cancer patients undergoing chemo(radio)- or immunotherapy treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven CRC stage IIB, III or IV or histologically or cytologically proven NSCLC stage III or IV
* Eligible and scheduled for first line chemotherapy, concurrent chemoradiotherapy or immunotherapy treatment with a planned duration of at least 12 weeks
* Performance status Eastern Cooperative Oncology Group (ECOG) score 0 or 1
* Age ≥ 18 years
* Written informed consent

Exclusion Criteria:

* Scheduled for first line chemotherapy, concurrent chemoradiotherapy or immunotherapy treatment starting ≤4 days after randomization
* Received radiotherapy within 2 months prior to the study
* Weight loss >10% in the last 6 months
* Body Mass Index < 20.0 kg/m2
* Life expectancy < 3 months
* Prescription of oral nutritional supplementation (ONS) before start of first line treatment based on hospital's standard practice
* Presence of ileostoma or ileal pouch
* Contra-indications to oral feeding, high protein nutrition or to the test product (including galactosaemia) in the opinion of the investigator
* Known pregnancy or lactation
* Current alcohol or drug abuse in the opinion of the investigator
* Investigator's uncertainty about the willingness or ability of the subject to comply with the protocol requirements
* Participation in any other studies involving investigational or marketed products concomitantly or within two weeks prior to entry into the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2019-01-17 (Actual); Primary Completion 2021-12-17 (Actual); Study Completion 2021-12-17 (Actual)

PRIMARY OUTCOMES:
The average protein intake (g/day and g/kg/day) corrected for baseline at the end of the first treatment cycle assessed with a 3-day food diary. | end of first treatment cycle (cycle length varies from 2-week, 3-week, 4-week or 6-weeks)
  The average protein intake (g/day and g/kg/day) corrected for baseline at the end of the first treatment cycle assessed with a 3-day food diary.

SECONDARY OUTCOMES:
Proportion of subjects with a protein intake above the lower limit of the ESPEN recommendations for protein intake | end of first treatment cycle (cycle length varies from 2-week, 3-week, 4-week or 6-weeks)
  Proportion of subjects with a protein intake above the lower limit of the ESPEN recommendations for protein intake
Change of body weight. | during 12 weeks (baseline till end of intervention at week 12]
  change of body weight measured with weighting scale

CONTACTS AND LOCATIONS:
Locations (14):
- Belgium (2):
  - UZ Gent, Ghent
  - AZ Nikolaas, Sint-Niklaas
- Estonia (2):
  - North Estonia Medical Centre, Tallinn
  - Tartu University Hospital, Tartu
- National Cancer Institute, Vilnius, Lithuania
- Netherlands (5):
  - Amphia Ziekenhuis, Breda
  - Maastricht University Medical Center, Maastricht
  - St. Antonius Hospital, Nieuwegein
  - Máxima Medisch Centrum, Veldhoven
  - Zaans Medisch Centrum, Zaandam
- Oslo University Hospital, Oslo, Norway
- Poland (2):
  - Szpital Kliniczny im. Heliodora Święcickiego UM w Poznaniu, Poznan
  - Hospital of Szczecin, Szczecin
- Centro Hospitalar Universitario Lisboa Norte EPE, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No